CLINICAL TRIAL: NCT06648122
Title: Association of Preoperative Inflammatory Markers With Preoperative Anxiety and Emergence Agitation in Children
Brief Title: Association of Inflammatory Markers With Preoperative Anxiety and Agitation
Status: Completed | Type: Observational
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Zehra Hatipoglu, MD, MD, Cukurova University
Other Study IDs: 09/2024;5
Record Dates: First submitted 2024-10-08; First posted 2024-10-18 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Preoperative Anxiety; Emergence Agitation
Keywords: Children; Preoperative anxiety; Emergence agitation; Inflammation
MeSH Terms: conditions — Emergence Delirium; Inflammation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: laboratory results — evaluation of laboratory results (hemogram results:WBC, RBC, Hematocrit, Monocyte count, Neutrophil count, Lymphocyte count, Platelet count, PDW, MPV, MLR, NLR, NMR, PLR, PMR, PNR, PWR, SII)

SUMMARY:
This study was planned as a prospective, observational study. The study will include pediatric patients aged 3-12 who will undergo surgery. Our hypothesis is that haemogram parameters, which are a simple, cheap and accessible method, and the inflammatory markers we obtain from them are associated with preoperative anxiety and emergence delirium

DETAILED DESCRIPTION:
Inclusion criteria for the study: Pediatric patients aged 5-12 years, in the ASA I-II groups, who will undergo surgery in ophthalmology, urological surgery, ENT surgery, pediatric surgery, orthopedic and plastic surgery. Exclusion criteria for the study can be listed as follows: Those with genetic diseases affecting brain development, those diagnosed with psychiatric and neurological diseases, patients with attention deficit, mental retardation, those with hematological and/or immune system disorders, patients who will undergo surgery in neurosurgery and cardiovascular surgery.

During the preoperative visit, parents and children will be informed and their written and verbal consent will be obtained. Patients will be taken to the preoperative waiting room and hemogram values and ratios (WBC, RBC, Hematocrit, Monocyte count, Neutrophil count, Lymphocyte count, Platelet count, PDW, MPV, MLR, NLR, NMR, PLR, PMR, PNR, PWR, SII) will be recorded from medical records. Demographic data (including age, gender, BMI, ASA score, fasting time, previous surgery, hospitalization status, the use of steroid), preoperative anxiety score (to be assessed with m-YPAS Turkish version), parental accompaniment, anxiety score of the parent (to be assessed with Likert scale), preoperative medication application, medications used in anesthesia, airway device, surgery and anesthesia durations will be recorded. The PAED score will be used for delirium agitation and all values will be recorded during the first 30 min. Pain scores (FLACC and VAS) will be recorded in the case report form.

ELIGIBILITY:
Inclusion criteria:

* Pediatric patients aged 5-12 years
* ASA I-II groups
* Pediatric patients who will undergo surgery in ophthalmology, urological surgery, ENT surgery, pediatric surgery, orthopedic and plastic surgery.

Exclusion criteria:

* Those with genetic disorders affecting brain development
* Those diagnosed with psychiatric and neurological diseases
* Patients with attention deficit, mental retardation
* Patients with hematological and/or immune system disorders
* Patients who will undergo surgery in neurosurgery and cardiovascular surgery.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children who will undergo surgery
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
PAED score | first 30 minutes in the postoperative unit.
  Emergence agitation will be evaluated in the postoperative unit with PAED scoring. PAED (Paediatric Emergence Delirium) parameters includes child makes eye contact with caregiver, child's actions are purposeful, child is aware of his/her surroundings, child is restless, child is inconsolable.All items are scored on a 0-4 point scale as occurring not at all, just a little, quite a bit, very much, If the sum of the five-parameter scale scores is ≥ 10, emergence agitation can be mentioned.

SECONDARY OUTCOMES:
mYPAS score | 15 minutes before surgery in the preoperative unit
  The Turkish version of the mYPAS (modified yale properative anxiety score) (Scores: min:23.3-max:100) scoring system will be used to assess preoperative anxiety in the preoperative unit. This score to be applied to each patient includes five categories and is applied observationally.
  The calculation of this score is as follows: (activity / 4 + emotional expression / 4 + the state of arousal / 4 + use of parents / 4 + vocalization / 6) × 100 / 5. Patients with m-YPAS≥40 will be considered anxious.
Demographic data | until the completion of surgery
  Age (year), gender, weight (kg) height (cm), BMI (kg/m2), previous surgery, fasting time, hospitalization state, parental accompaniment, score of the parent anxiety (to be assessed with Likert scale), preoperative medication application, drugs used in anesthesia, surgery and anesthesia durations, pain scores will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Faculty of Medicine, Department of Anesthesiology, Adana, Turkey, Turkey (Türkiye)